CLINICAL TRIAL: NCT05557916
Title: A Randomised Control Trial of Rehabilitation With or Without a Knee Orthosis Following Meniscal Repair
Brief Title: Rehabilitation With or Without Knee Orthosis Following Meniscal Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anders Stalman, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Meniscal suture orthosis study
Record Dates: First submitted 2022-02-20; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Meniscal Tear

STUDY DESIGN:
Intervention Model Description: Randomised control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard rehab group (Active Comparator): This group will follow the clinics standard rehab protocol, wherein they have a knee orthosis for six weeks, with flexion limited to 0-30 degress week 0-2, 0-60 degrees week 2-4 and 0-90 degrees week 4-6. Crouching is not permitted week 6-12.
  Interventions: Other: Standard rehab
- Accelerated rehab group (Active Comparator): accelerated rehab group, wherein they are permitted to perform range of motion training within their comfort zone. Running is permitted after 8 weeks, contact sports 4 months postoperatively
  Interventions: Other: accelerated rehab group

INTERVENTIONS:
Other: Standard rehab — Standard rehab protocol including knee orthosis following meniscal repair
  Arms: Standard rehab group
Other: accelerated rehab group — accelerated rehab group, no orthosis
  Arms: Accelerated rehab group

SUMMARY:
RCT to determine if a less restrictive postoperative rehabilitation protocol following meniscal repair results in a faster return to normal knee function without compromising rates of healing.

DETAILED DESCRIPTION:
The purpose of the study is to compare rehabilitation after meniscal repair with or without the use of a knee orthosis. There is conflicting evidence regarding optimal postoperative rehabilitation following meniscal repair with ACLR. Many surgeons advocate the use of a knee orthosis which restricts flexion during the first 4-6 weeks following surgery. Some also avoid weight baring and crouching for various periods of time. This is due to the perceived risk that the healing meniscus is exposed to unnecessary strain, potentially compromising healing. There is however evidence that fewer postoperative restriction in the setting of meniscal repair in conjunction with ACLR does not compromise meniscal healing. There is also evidence that accelerated rehabilitation following isolated meniscal repair does not increase the risk of failure.

The study design is a prospective randomized study with equal groups.

A power analysis has been performed indicating that 57 patients in each group are required to detect a significant difference between groups, as such a cohort of 120 patients will be recruited. Randomisation will continue until 60 patients are allocated to both groups.

Randomization process and study design will be done according to the CONSORT guidelines.

ELIGIBILITY:
Inclusion Criteria:

• Meniscal tear in the peripheral zone of the meniscus, repaired using at least two sutures.

Exclusion Criteria:

* Associated injury of the knee requiring surgical or non-surgical intervention that precludes the patient from completing accelerated rehabilitation- fracture, concomitant ligament or cartilage injury.
* Previous meniscal repair in the affected meniscus
* BMI over 30

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Biodex isokinetic quadriceps strength at 6 months | six months
  Patients will undergo Biodex Isokinetic measurement at 6 months

SECONDARY OUTCOMES:
Rates of failure | two years
  Rates of failure, defined as reoperation with meniscal resection within two years of the repair.
Knee injury and Osteoarthritis Outcome Score (KOOS) | preoperative, six months, two years
  Patients will complete the KOOS at specific time points to evaluate subjective knee function throughout treatment. Score range from 0 to 100, with higher scores indicating better results
Change from baseline Biodex isokinetic quadriceps strength at 24 months | 2 years
  Patients will undergo Biodex Isokinetic measurement at 24 months
Goniometric measurement: Knee flexion and extension | 2 weeks, 6 weeks, 6 months, 2 years
  Patients will undergo Goniometric measurement at specific time points to evaluate knee range of motion
IKDC | Pre-operative, 6 months, 2 years
  Patients will complete the IKDC at specific time points to evaluate subjective knee function throughout treatment. Score range from 0 to 100, with higher scores indicating better results
Tegner activity score | Pre-operative, 6 months, 2 years
  Patients will complete the Tegner activity score at specific time points to evaluate Activity in sports throughout treatment, Assesses activity level with specific emphasis on knee; scores range from 1 (least strenuous activity) to 10 (high knee demanding activity on professional sports level)
Lysholm score | Pre-operative, 6 months, 2 years
  Patients will complete the Lysholm score at specific time points to evaluate subjective knee function throughout treatment. Score range from 0 to 100, with higher scores indicating better results
Measurement of circumference of the knee | Pre-operative, 6 weeks, 3 months, 6 months, 2 years
  Circumference of the knee will be measured at mid-patella and 15cm above superior border of patella. They will be compared with contralateral knee to compare swelling.
Functional knee tests | 6 weeks, 6 months, 2 years
  patients will undergo functional knee tests (ie Single hop test for difference, 30s chair-stand test

CONTACTS AND LOCATIONS:
Overall Officials: Erik Rönnblad, Study Director — Centrum för idrottsforskning och utbildning (CIFU) Adress: Valhallavägen 91, 11427 Stockholm
Locations (2):
- Sweden (2):
  - Centrum för idrottsforskning och utbildning (CIFU), Stockholm
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No